CLINICAL TRIAL: NCT02940275
Title: Population Research of Sublingual Microcirculation Data of Patients With Systemic Diseases
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201609021RINB
Record Dates: First submitted 2016-10-18; First posted 2016-10-20 (Estimated); Last update posted 2019-03-04 (Actual); Status verified 2019-02

CONDITIONS: Hypertension; Diabetes Mellitus
MeSH Terms: conditions — Hypertension; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- Hypertension
- Diabetes mellitus
- Hypertension and diabetes mellitus
- End stage kidney disease
- Kidney transplant recipient
- Coronary artery disease
- Peripheral arterial occlusive disease

SUMMARY:
This is an observational clinical study, patients with systemic diseases will be enrolled according to the inclusion and exclusion criteria. Patients will received the examination of sublingual microcirculation by using incident dark field video microscope (Cytocam，Braedius Battery Powered Transilluminator). The microcirculation data includes total small vessel density, perfused small vessel density, microvascular flow index, and heterogeneity index. The patients will be divided into right groups according to their systemic diseases as follows: group 1 hypertension (60 patients), group 2 diabetes mellitus (60), group 3 hypertension and diabetes mellitus (60), group 4 end stage renal disease with hemodialysis (60), group 5 kidney transplant recipients (60), group 6 coronary artery disease (60), and group 7 peripheral arterial occlusive disease (60).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 20 to 79 years old
* BMI ranged from 18.5 to 27 kg/m2
* Presence of one of the condition

  * Diagnosed hypertension > 6 months, without other systemic diseases
  * Diagnosed diabetes mellitus > 6 months, without other systemic diseases
  * Diagnosed with both hypertension and diabetes mellitus > 6 months, without other systemic diseases
  * Diagnosed with end stage renal disease > 6 months
  * Received renal replacement therapy > 6 months
  * Diagnosed with coronary artery disease > 6 months
  * Diagnosed with peripheral arterial occlusive diseases > 6 months

Exclusion Criteria:

* Diagnosed with sepsis, major trauma, or admission to ICU within one month
* Body temperature higher than 37.5 ℃ or lower than 35.5 ℃
* Any on of the following condition
* Asthma
* Chronic obstructive pulmonary disease
* Endocrine diseases
* Hematological disorders
* Uncured cancer
* Chronic uncured infection
* Other major disease with limited daily activity
* Non-native speakers

Ages: 20 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with systemic diseases
Sampling Method: Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2016-10-17; Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Perfused small vessel density of sublingual small vessels measured by Cytocam | Once at enrollment

SECONDARY OUTCOMES:
Total small vessel density of sublingual small vessels measured by Cytocam | Once at enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan